CLINICAL TRIAL: NCT03808155
Title: Prevention of Postoperative Urinary Retention With Treatment of Tamsulosin 5 Days Prior to Lower Limb Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kantonsspital Graubünden (Other)
Responsible Party: Principal Investigator, PD Dr. med. Räto T. Strebel, Head of Urology, Kantonsspital Graubünden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GR20192021
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-10

CONDITIONS: Urinary Retention Postoperative; Arthropathy of Knee; Arthropathy of Hip
Keywords: Urinary retention; Tamsulosin
MeSH Terms: conditions — Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin (Active Comparator): The study specific product Tamsulosin 0.4mg, a tablet which is taken once a day per os five days prior to the operation and two days after the operation.
  Interventions: Drug: Tamsulosin
- Placebo Oral Tablet (Placebo Comparator): The placebo is taken once a day per os five days prior to the operation and two days after the operation.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tamsulosin — The drug ist taken once a day per os five days prior to the operation and two days after the operation.
  Other Names: Pradif
  Arms: Tamsulosin
Drug: Placebo Oral Tablet — The placebo ist taken once a day per os five days prior to the operation and two days after the operation.
  Arms: Placebo Oral Tablet

SUMMARY:
Various studies have shown that the risk of suffering a urinary retention after knee or hip prosthesis surgery is 10-80%. The aim of the study is to reduce this riks. For this purpose, it is investigated whether a previously known drug (tamsulosin) which is used in bladder emptying disorders, can achieve a reduction in urinary retention after surgery. After the patients agree to participate in the study, they are examined in our urological clinic. Uroflowmetry is performed with sonographic residual volume measurement and prostate volume measurement. Furthermore, a standardized Voiding questionaire (IPSS) is completed. This study is conducted as a double-blind study using a placebo control group. The drug / placebo is taken once a day, five days before and two days after surgery. Subsequently, it is observed whether it comes to a urinary retention or not. After the operation, no further urological checks are planned or needed.

DETAILED DESCRIPTION:
Study Category and rationale:

This study uses a well-known drug (tamsulosin) which is authorised in Switzerland and widely used to treat obstructive voiding problems. In our case the indication is different from that specified in the prescribing information, but it is within the same disease group, which in our case is to prevent urinary retention. Therefore according to the legal ordinance on clinical trials (ClinO), this study is classified as a clinical trial, research with collection of health-related personal data and placebo controlled of the category B.

Objective:

Our goal is to reduce the rate of postoperative urinary retention after lower limb arthroplasty. For this purpose, we plan to investigate whether an already known drug (Tamsulosin), which is widely used for bladder emptying disorders, could reduce the rate of postoperative urinary retention.

Outcomes:

The primary outcome is the occurrence of urinary retention during the 48 postoperative hours. The secondary outcome is the influence of other clinical factors on the occurrence of urinary retention as type of anaesthesia, preoperative residual volume, prostate size and international prostate symptom score (IPSS).

Measurement and procedures:

Once the decision for lower limb arthroplasty is made during the planned orthopaedic consultation, the patient will receive a participant information sheet and the informed consent. If the patient is interested to take part in the study he will receive an appointment in the urological clinic at least six days before the operation. During the appointment a urological specialist will explain the entire study. A uroflowmetry with sonographic measurement of residual volume and prostate volume will be performed. Furthermore, the patient will fill out an IPSS-questionnaire. After the appointment the drug/placebo will be handed out to the patient, which should be taken once a day five days prior to the operation, on the day of surgery and two days thereafter.

Study product:

The study specific product Tamsulosin 0.4mg, a tablet which is taken once a day per os five days prior to the operation and two days after the operation.

Control intervention:

Placebo.

Number of participants with rationale:

The number of participants projected for the entire study is 170. Thus 85 patients in the drug-treatment group and 85 patients for the placebo-treatment group.

ELIGIBILITY:
Inclusion Criteria:

- male adults undergoing elective hip- or knee arthroplasty

Exclusion Criteria:

* women
* underage patients
* pre-existing treatment with tamsulosin or other prostate affecting medication
* patients who underwent transurethral resection of the prostate or prostatectomy
* patients with urethral strictures
* patients with neurological bladder dysfunction
* Known allergy to tamsulosin
* Hypotensive disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The participant has to be a genectic male with all male organs.
Enrollment: 170 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of urinary retention | 48 hours postoperatively
  The primary outcome is the occurrence of urinary retention during the 48 postoperative hours.

SECONDARY OUTCOMES:
Type of anaesthesia | 48 hours postoperatively
  Did the patient undergo general anaesthesia, spinal anaesthesia or regional anaesthesia
Preoperative residual volume | Minimum 6 days before the planned operation.
  Preoperatively the residual volume will be measured in milliliters (mL) by ultrasound.
Prostate size | Minimum 6 days before the planned operation.
  Preoperatively the prostate volume will be measured in milliliters (mL) by ultrasound.
International prostate symptom score (IPSS). | Minimum 6 days before the planned operation.
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).

CONTACTS AND LOCATIONS:
Overall Officials: Räto T. Strebel, PD Dr. med., Principal Investigator — Kantonsspital Graubünden
Locations (1):
- Kantonsspital Graubünden, Chur, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No